CLINICAL TRIAL: NCT06700239
Title: The STTAR-US Study: A Pivotal Study of Transcatheter Tricuspid Annular Repair in the US
Acronym: STTAR-US
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Micro Interventional Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MID-004
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Tricuspid Regurgitation Functional; Tricuspid Regurgitation; Severe Tricuspid Valve Regurgitation
Keywords: MIA-T; severe TR; severe functional TR
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Two cohorts One (1) cohort will randomize subjects at a 1:1 ratio against commercially available TEER Device (control group).
  One (1) cohort is a single arm cohort for patients deemed unfavorable for TEER and the local heart team determines the patient is not optimal for valve replacement.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Randomized Cohort TEER (Active Comparator): MIA-T vs. TEER
  Interventions: Device: MIA_T Device
- Single Arm Cohort (Experimental): MIA-T
  Interventions: Device: MIA_T Device
- Roll-in (Experimental): MIA-T device for physicians training prior to initiating randomized cohort enrollment.
  Interventions: Device: MIA_T Device

INTERVENTIONS:
Device: MIA_T Device — MIA-T Device

SUMMARY:
Purpose of this clinical study is to demonstrate the safety and efficacy of MIA-T system in improving clinical outcomes in symptomatic patients with severe tricuspid regurgitation (TR grade ≥3) despite optimal medical therapy, who have been determined by the site's local heart team to be at intermediate or greater estimated risk for mortality and morbidity with tricuspid valve surgery.

DETAILED DESCRIPTION:
A prospective, multi-center, randomized, controlled, pivotal study of the MIA Percutaneous Tricuspid Annuloplasty System (MIA-T) in symptomatic subjects with severe (≥3) TR despite optimal medical therapy.

The study will randomize eligible subjects in two (2) cohorts at up to 40 sites.

ELIGIBILITY:
Inclusion Criteria:

* Subject has severe functional TR (≥ 3). Note: If any cardiac procedure(s) occur after eligibility was determined, TR severity will need to be re-assessed 30 days after any cardiac procedure(s)
* In the judgment of the site's local heart team patient is at intermediate or greater risk for morbidity & mortality with tricuspid valve surgery, and has been adequately treated per applicable standards with optimized medical therapy for the treatment of TR (e.g. diuretics) and stable for at least 30 days prior to enrollment.
* New York Heart Association (NYHA) Functional Class II, III or ambulatory class IV

Exclusion Criteria:

* Systolic pulmonary artery pressure (sPAP) > 70 mmHg or > 5 wood units (WU) despite vasodilator therapy
* Severe uncontrolled hypertension Systolic Blood Pressure (SBP) ≥ 180 mmHg and/or Diastolic Blood Pressure (DBP) ≥ 110 mm Hg
* Previous tricuspid valve repair or replacement (transcatheter or surgical approach)
* Subjects with concomitant left-sided valve disease will have the option of receiving a left-sided intervention (e.g. TMVR or TAVR) and waiting 60 days prior to being reassessed for the study
* Myocardial infarction (MI), known unstable angina, symptomatic coronary artery disease (CAD) where revascularization is possible within 60 days prior to enrollment
* Anatomy that precludes safe placement of anchors around the annulus
* Hemodynamic instability defined as systolic pressure < 90 mmHg requiring pressor support within the last 30 days

Echo Criteria -

* Subject has severe functional TR (determined by the ICL). Note: If any cardiac procedure(s) occur after eligibility was determined, TR severity will need to be re-assessed 30 days after any cardiac procedure(s)
* No presence of Cardiac Implantable Electronic Devices (CIED) leads causing the TR
* No significant annular calcification
* Left Ventricular Ejection Fraction (LVEF) ≥ 20%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | 12 months
  Composite endpoint of the following components:
  * All-cause mortality
  * Tricuspid valve intervention (percutaneous or surgery)
  * Heart Failure Hospitalization
Primary Safety Endpoint | 30 days
  Freedom from MAE, including:
  * Cardiovascular mortality
  * New Onset Renal Failure
  * Endocarditis requiring surgery
  * Non-elective cardiovascular surgery for device-related AE post-index procedure

SECONDARY OUTCOMES:
Freedom from all-cause mortality at all study timepoints | 1Month, 6Month, 12Month, 2Years, 3Years, 4Years, and 5Years
Freedom from heart failure hospitalizations at all study timepoints | 1Month, 6Month, 12Month, 2Years, 3Years, 4Years, and 5Years
Clinical Success Rate | 1Month
Intraprocedural Success Rate | 1Month
Freedom from Major Adverse Events (MAE) at all study time points. | 1Month, 6Month, 12Month, 2Years, 3Years, 4Years, and 5Years
Prevalence of Device or Procedure-Related Adverse Events (AE) | 1Month, 6Month, 12Month, 2Years, 3Years, 4Years, and 5Years
Core Lab assessment of change in other pertinent echo | 1Month, 6Month, 12Month, 2Years, 3Years, 4Years, and 5Years
Change in NT-proBNP | 1Month, 6Month, 12Month, 2Years, 3Years, 4Years, and 5Years
Change in gamma-GTP | 1Month, 6Month, 12Month, 2Years, 3Years, 4Years, and 5Years
Change in eGFR | 1Month, 6Month, 12Month, 2Years, 3Years, 4Years, and 5Years
Change in MELD score (liver function) | 1Month, 6Month, 12Month, 2Years, 3Years, 4Years, and 5Years
Change in SF-36 QoL scores | 1Month, 6Month, 12Month, 2Years, 3Years, 4Years, and 5Years

OTHER OUTCOMES:
TR Grade Reduction | 12 months
  Change in TR grade to moderate or less
KCCQ Reduction | 12 months
  Average change in patients overall KCCQ summary scores by ≥ 10

IPD SHARING:
Plan to Share IPD: No